CLINICAL TRIAL: NCT02498379
Title: PET-Magnetic Resonance (MR) Imaging of Natriuretic Peptide Receptor C (NPR-C) in Carotid Atherosclerosis With [64]Cu-25%CANF-Comb (Volunteer - BioDistribution and Safety Study)
Brief Title: PET Imaging of Natriuretic Peptide Receptor C (NPR-C) in Carotid Atherosclerosis (Volunteer - BioD and Safety Study)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Pamela Woodard, MD, Sponsor-Investigator, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201409006V
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Atherosclerosis
Keywords: novel radiotracer; biodistribution; safety
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cu[64]-25%CANF-Comb (Experimental): Single IV injection of 4-8 mCi Cu[64]-25%CANF-Comb followed by PET-CT scan at 1-4 hours, 5-10 hours, and 22-26 hours or 46-50 hours post injection.
  Interventions: Drug: Cu[64]-25%CANF-Comb

INTERVENTIONS:
Drug: Cu[64]-25%CANF-Comb — Intravenous injection of 4-8 mCi of Cu[64]-25%CANF-Comb with PET-CT scans performed 1-4 hours, 5-10 hours, and 22-26 hours or 46-50 hours after injection.

SUMMARY:
This study is designed to assess the safety, biodistribution and dosimetry of the novel atherosclerotic imaging PET radiotracer, Cu[64]-25%-CANF-Comb.

DETAILED DESCRIPTION:
This study is a single center, open-label baseline controlled imaging study designed to demonstrate safety, biodistribution and dosimetry of the radiopharmaceutical Cu[64]-25%CANF-Comb (Cu = copper; CANF = C-type Atrial Natriuretic Factor) in healthy, adult volunteers. By definition a "healthy" volunteer is an individual who, by physical exam and baseline electrocardiogram, has no evidence of cardiovascular disease and, by history, is not under the care of a physician for any active medical conditions.

Each volunteer will receive a single intravenous bolus injection of 4-8 mCi of the investigational radiotracer Cu[64]-25%CANF-Comb followed by whole body static PET-CT imaging at 3 of 4 dedicated imaging time points, (1-4 hours, 5-10 hours, and 22-26 hours or 46-50 hours post injection). For safety assessment, a physical examination will be performed at baseline and at the completion of all imaging to assess for interval change. An EKG and vital signs will be obtained baseline, at each imaging time point to assess for interval change. Blood will be drawn at baseline, and at each imaging time point to assess for interval change in serum chemistries and complete blood count. Urine will be collected at baseline and at each imaging time point to assess for interval change in urinalysis results.

The amount of radioactive tracer in the blood and urine will also be assessed on all 8 adult normal volunteer subjects. One-mL blood samples will be obtained at baseline, 1, 2, 4, and 24 hours post Cu[64]-25%CANF-Comb injection and prior to discharge. Urine will be collected as a single accumulated collection over 24 hours immediately following injection of Cu[64]-25%CANF-Comb and prior to discharge.

Tracer biodistribution will be evaluated by measuring tracer uptake in various organs in the torso on the PET-CT scan. The organs used to describe the biodistribution of the radiopharmaceutical will be blood, liver, kidneys, spleen, heart, bone, muscle and other organs showing significant uptake. Only organs and tissues containing a visible accumulation of activity will be selected for image quantification. Region of Interests (ROIs) will be drawn to measure average activity concentration in each organ or tissue. Values in three-dimensional region of interest (3D-ROI) traced on the contour of the organs will be used. For the large organs such as the liver, a large elliptical ROI encompassing as much of the organ as possible will be used to obtain an average pixel value. To estimate bone activity, a narrow, irregular ROIs will be drawn to approximate the visible cross section of the ilium or large vertebrae, and the average pixel value will be used. For blood activity, the average pixel intensity in a large 3D-ROI drawn over the left ventricle will be used, thereby avoiding partial volume effects. Muscle activity will be taken as the average value in a large elliptical ROI in the region of the buttocks as seen on MR images. Fat activity will be taken as the average value in a large elliptical ROI in the region of the subcutaneous abdominal fat. All other non-listed organ's activity concentration will be measured in a similar fashion.

Residence times will be calculated by analytical integration of the fitted time taking into account the radioactive decay of Cu[64]. Residence times will be expressed in hours and normalized to one unit injected activity. Blood activity will be also assigned to the heart, lungs and bone marrow, organs for which activity will be not measured directly with an ROI. The heart and lungs will be assigned a blood fraction based on their respective blood volumes. Activity measured in bone is assigned half to cancellous bone and half to cortical bone.

The percent injected dose values will be calculated by extrapolating the measured activity concentration in each organ to the whole organ using standard organ and tissue volumes. These standard volumes will be normalized to each patient's weight. Time activity curves will be then constructed from these values for all organs for which ROIs were drawn including liver, spleen, kidneys, bone, muscle blood pool and remainder of body by combining the data from all the patients. The blood content of each organ will be included with the organ where possible rather than assigning it uniformly to the remainder of body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (4 men and 4 women)
* No evidence of cardiovascular disease and not under care of a physician for any active medical condition
* Health status confirmed by physical exam and ECG
* Signed informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Inability to lie still for up to 60 min with arms above head for PET-CT imaging
* Unwilling to comply with study procedures and unavailable for the duration of the study.
* Inability to provide written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Biodistribution, dosimetry and safety of Cu[64]-25%CANF-Comb in normal healthy adult volunteers. | 24-48 hours
  Biodistribution by PET-CT (Cu[64]-25%CANF-Comb uptake in blood, liver, kidneys, spleen, heart, bone, muscle); Amount of radioactive tracer in the blood and urine; Difference in physical examination findings, vital signs, serum and urine laboratory values and EKG results from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Woodard, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St.Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu Y, Pressly ED, Abendschein DR, Hawker CJ, Woodard GE, Woodard PK, Welch MJ. Targeting angiogenesis using a C-type atrial natriuretic factor-conjugated nanoprobe and PET. J Nucl Med. 2011 Dec;52(12):1956-63. doi: 10.2967/jnumed.111.089581. Epub 2011 Nov 2. PMID 22049461
- [Background] Liu Y, Abendschein D, Woodard GE, Rossin R, McCommis K, Zheng J, Welch MJ, Woodard PK. Molecular imaging of atherosclerotic plaque with (64)Cu-labeled natriuretic peptide and PET. J Nucl Med. 2010 Jan;51(1):85-91. doi: 10.2967/jnumed.109.066977. Epub 2009 Dec 15. PMID 20008978